CLINICAL TRIAL: NCT06477614
Title: Anti-cancer DC Cell Vaccination to Treat Advanced Solid Tumors: Phase I Clinical Trial
Brief Title: Anti-cancer DC Cell Vaccination to Treat Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZVACCINE-DC-022
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult; DC
Keywords: Solid Tumor; DC Vaccine; gp96

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placental gp96 induced DC cell Vaccine (Experimental)
  Interventions: Biological: DC cell Vaccine
- Tumor-derived gp96 induced DC cell Vaccine (Experimental)
  Interventions: Biological: DC cell Vaccine

INTERVENTIONS:
Biological: DC cell Vaccine — Deliver DC cell vaccine into patients for anti-ancer therapy.

SUMMARY:
Placental or tumor-derived heat shock protein gp96 is collected, purified, and stored. The DC cells are isolated from the patient's blood and then cocultured with the gp96 to obtain the activated DC cell product. The manufactured DC cells are subcutaneously or intra-tumor injected into the patient. Clinical studies will be performed to test anti-cancer function of the DC vaccination for immunotherapy of cancer patients. In this phase I study, the safety, tolerance, and preliminary efficacy of the DC vaccine immunotherapy on advanced cancers will firstly be evaluated.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced solid cancers, with written consent for this study;
2. Perform biopsy to get fresh sample for generation gp96 protein; Collect DC cells from the cancer patient;
3. Produce appropriate DC cell vaccine and deliver the vaccine into selected patients via local injections, and follow up closely to collect related results as required;
4. To enhance the killing capability, cotreatment the patients with vaccine aduvants or PD1/PDL1/CTLA4 antibodies may be applied;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer; 2. Life expectancy >12 weeks; 3. Adequate heart, lung, liver, kidney, and blood function; 4. Available high quality vaccine for human use; 5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

-

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV, HCV, HIV, et al;
3. Known HIV positivity;
4. Active infectious disease related to bacteria, virus,fungi,et al;
5. Other severe diseases that the investigators consider not appropriate;
6. Pregnant or lactating women;
7. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
8. Other conditions that the investigators consider not appropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | Six months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the vaccine, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | Six months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China